CLINICAL TRIAL: NCT04468711
Title: The Impact of Vitamin D Supplementation as an Adjuvant Therapy on Clinical Outcome in Patients With Severe Atopic Dermatitis
Brief Title: Vitamin D in Egyptian Children With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Noha Mansour, Principal Investigator, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-2018
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): vitamin D plus topical 1% hydrocortisone cream twice daily
  Interventions: Drug: Vitamin D
- placebo group (Placebo Comparator): placebo plus plus topical 1% hydrocortisone cream twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Vitamin D plus topical 1% hydrocortisone cream twice daily
  Other Names: plus topical 1% hydrocortisone cream twice daily
  Arms: treatment group
Drug: Placebo — placebo plus topical 1% hydrocortisone cream twice daily
  Arms: placebo group

SUMMARY:
There is an emergent evidence demonstrating the role of Vitamin D deficiency in eczema. Vitamin D supplementation with standard treatment yielded positive clinical outcomes for children and adolescents with mild and moderate AD; however, the potential benefit of vitamin D in severe cases remains unclear

ELIGIBILITY:
Inclusion Criteria:

1.diagnosis of severe AD according to Hanifin and Rajka criteria and the Eczema Area and Severity Index (EASI) score

Exclusion Criteria:

1. serious skin disorder other than AD.
2. taking systemic corticosteroids or anti-inflammatory medications, prior vitamin D supplementation
3. receiving oral or topical antibiotics or topical calcineurin inhibitors for at least one week prior to enrollment
4. known gut absorption problem, presence of active skin infection at baseline any known hepatic and/or renal disease.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
difference in the mean Eczema Area and Severity Index (EASI) score at the end of the study | 12 weeks
the average percent change in Eczema Area and Severity Index (EASI) score at the end of the study | 12 weeks

SECONDARY OUTCOMES:
Difference in proportion of patients with a reduction from baseline of 75 % in Eczema Area and Severity Index (EASI) score | 12 weeks
  EASI 75
Difference in proportion of patients with a reduction from baseline of (50 or more up to 75) in Eczema Area and Severity Index (EASI) score | 12 weeks
  EASI 50
Difference in proportion of patients with a reduction from baseline of <50 n Eczema Area and Severity Index (EASI) score | 12 weeks
  EASI<50

CONTACTS AND LOCATIONS:
Locations (1):
- NHTRMI, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No